CLINICAL TRIAL: NCT02377635
Title: Selenium and Arsenic Pharmacodynamics
Acronym: SEASP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: University of Chicago (Other); University of Calgary (Other); University of Alberta (Other); Emory University (Other); Wagner College, Staten Island, NY, USA (Unknown); Applied Speciation and Consulting LLC, WA, USA (Unknown)
Responsible Party: Principal Investigator, Graham George, Ph.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 14-284; Grand Challenges Canada/7315 (Other Grant/Funding Number: Government of Canada)
Record Dates: First submitted 2015-02-10; First posted 2015-03-03 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Arsenic Poisoning Chronic
Keywords: Arsenic; Arsenicosis
MeSH Terms: interventions — Sodium Chloride; Sodium Chloride, Dietary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Drug: Anhydrous selenite (Se-77), single dose 0.8mg, orally administered as a 100 ml purified water solution
  Interventions: Dietary Supplement: Anhydrous selenite
- Control (Placebo Comparator): Drug: Placebo sodium chloride (table salt), orally administered as a 100 ml purified water solution
  Interventions: Dietary Supplement: Sodium chloride

INTERVENTIONS:
Dietary Supplement: Anhydrous selenite — 40 volunteer sufferers will be housed in a local private in-patient clinic where they will follow a fixed, communal diet consisting of drinking water and meals from their village. On a 6th day we will give a single dose of placebo (sodium chloride) or anhydrous sodium selenite (0.8mg selenium) labelled with a non-radioactive naturally occurring isotope (77Se), to distinguish it from selenium already in the body.
  Other Names: Sodium selenite anhydrous
  Arms: Treatment
Dietary Supplement: Sodium chloride — 40 volunteer sufferers will be housed in a local private in-patient clinic where they will follow a fixed, communal diet consisting of drinking water and meals from their village. On a 6th day we will give a single dose of placebo (sodium chloride) or anhydrous sodium selenite (0.8mg selenium) labelled with a non-radioactive naturally occurring isotope (77Se), to distinguish it from selenium already in the body.
  Other Names: Table salt
  Arms: Control

SUMMARY:
This clinical trial should prove that selenium can treat arsenic exposure in humans by promoting excretion. The new trial differs from previous trials in that participants will be maintained in a local clinic and provided with food and water from their home villages. The purpose of this study to determine the fate of selenium supplements in feces, urine and blood of volunteers living in conditions of high arsenic load in drinking water. The use of a clinic will enable monitoring of all intake and excretion of both arsenic and selenium, and will ensure that participants take their selenium doses or placebo as appropriate. This proof of concept is absolutely essential groundwork for any remediation strategy involving selenium supplements.

DETAILED DESCRIPTION:
Main Purpose:

Determine the fate of selenium supplements in feces, urine and blood through a new Phase I/II clinical trial pharmacodynamics study in Bangladesh. This will include conventional analysis of feces, urine and blood samples, tracing the fate of selenium by administering isotopically enriched 77Se (a naturally occurring non-radioactive stable isotope). The use of 77Se will allow us to discriminate between endogenous selenium already in the bodies of the trial participants (patients) from the administered selenium given to the patients.

Clinical Trial Hypotheses:

* In a group of patients exhibiting symptoms of arsenicosis (chronic low-level arsenic poisoning), a single, elevated dose of anhydrous sodium selenite leads to excretion of arsenic at levels significantly higher than patients receiving placebo.
* In the selenite-supplemented (treatment) group, the total arsenic excreted is significantly higher than that consumed in the diet and drinking water.
* In the treatment group, selenium co-excreting with arsenic originates from the administered selenium supplement, rather than from endogenous selenium.
* The ratio of arsenic to selenium in the feces, urine and blood of the treatment group following administration of the selenium supplement is approximately 1:1, consistent with the formation of the discrete molecular entity, the seleno bis-S-glutathionyl arsinium anion discovered in the investigators' earlier animal experiments.

The process to be followed:

A tightly controlled Phase I/II clinical trial in Bangladesh to prove that selenium can remove arsenic from victims' bodies. 40 volunteer arsenicosis sufferers will be housed in a local private in-patient clinic for 10 consecutive days. While in the clinic, they will follow a fixed, communal diet consisting of drinking water and meals from their village. On the 6th day in the clinic investigators will give a single dose of either placebo (table salt, 0.8 mg) or anhydrous sodium selenite (0.8 mg selenium) labelled with a non-radioactive naturally occurring isotope (77Se), to distinguish it from selenium already in the body. Placebo and anhydrous sodium selenite look similar and taste very much alike. Placebo or anhydrous sodium selenite will be supplied in a powdered form at the bottom of a glass and diluted by 100 ml of purified water immediately before being ingested by participants under close control by the clinical staff. The investigators will analyze arsenic and selenium levels in feces, urine and blood samples before and after the dose, and will use molecular speciation analyses to determine their chemical form in blood, urine and feces. Also, investigators will analyze arsenic and selenium levels in finger- and toenails and hair at the beginning of the trial as a possible biomarker of As exposure.

ELIGIBILITY:
Inclusion Criteria:

The participants in this study are

1. healthy adult (18-65 years of age) male Bangladeshi volunteers from Laksam Upazila,
2. who are exposed to arsenic through their normal source of drinking water;
3. who are otherwise healthy except that show some signs of chronic arsenic toxicity (arsenicosis);
4. have not consumed selenium-containing supplements with last 6 months;
5. not concurrently participating or have participated in any other clinical trial within at least 30 days of registration to the current trial.

Exclusion Criteria:

1. Recent history of consuming selenium, concurrent participation or recent participation in any other clinical trial within at least 30 days of registration to the current trial, and people who recently moved in the area.
2. Prior clinical trial, recruits will undertake a medical examination by physician. Since chronic kidney disease and alcoholic and viral cirrhosis are common in rural Bangladesh and both conditions might impact selenium and arsenic metabolism, recruits will also be screened through a baseline CMP (Comprehensive Metabolic Panel) , CBC (Complete Blood Count), and INR (International Normalized Ratio of Prothrombin Time as Liver Function Test) panel. Evidence or history of significant hematologic, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, musculoskeletal, immunologic, neurologic or dermatologic disease (including drug allergies that are clinically significant) which, by opinion of investigators, could pose a risk to the safety of the individual or the valid conduct of the study will exclude recruits from the participation.
3. Current evidence of or history of cancer; evidence of hepatitis B, hepatitis C, human immunodeficiency virus (HIV) infection upon serological testing; evidence of active communicable disease or febrile illness (e.g., bronchopulmonary, urinary or gastrointestinal) within 7 days prior to study will exclude recruits from participation.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02-10; Primary Completion 2016-12-19 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
Blood As and Se concentrations and chemistry | 10 days
  The ICPMS technique will be used to analyze arsenic and selenium levels in blood samples before and after the dose. The molecular speciation analyses (IC-ICP-MS) will be applied to determine their chemical form in blood.
Urinary As and Se concentrations and chemistry | 10 days
  The ICPMS technique will be used to analyze arsenic and selenium levels in urine samples before and after the dose. The molecular speciation analyses (IC-ICP-MS) will be applied to determine their chemical form in urine.
Fecal As and Se concentrations and chemistry | 10 days
  The ICPMS technique will be used to analyze arsenic and selenium levels in feces samples before and after the dose. The molecular speciation analyses (IC-ICP-MS) will be applied to determine their chemical form in feces.

SECONDARY OUTCOMES:
The absolute concentrations of 77Se and the ratios (total Se/77Se) and (As/77Se) determined in blood, at each time point of the study. | 10 days
  Quantitative analysis (ICP-MS) of As, 77Se and total Se to evaluate the effect of Se supplementation on binding and excretion of arsenic as opposed to the mobilization of endogenous Se in a body.
The absolute concentrations of 77Se and the ratios (total Se/77Se) and (As/77Se) determined in urine, at each time point of the study. | 10 days
  Quantitative analysis (ICP-MS) of As, 77Se and total Se to evaluate the effect of Quantitative analysis (ICP-MS) of As, 77Se and total Se to evaluate the effect of Se supplementation on excretion of arsenic as opposed to the mobilization of endogenous Se in a body.
The absolute concentrations of 77Se and the ratios (total Se/77Se) and (As/77Se) determined in feces, at each time point of the study. | 10 days
  Quantitative analysis (ICP-MS) of As, 77Se and total Se to evaluate the effect of Se supplementation on excretion of arsenic as opposed to the mobilization of endogenous Se in a body.
Arsenic and selenium concentrations in hair, finger- and toenails | 1 day
  Quantitative analysis (ICP-MS) of As and Se content in keratinous tissues as a possible biomarker of As exposure

CONTACTS AND LOCATIONS:
Overall Officials: Graham N George, D.Phil., Principal Investigator — University of Saskatchewan
Locations (1):
- Unity Hospital Pvt LTD, Lākshām, Comilla, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gailer J, George GN, Pickering IJ, Prince RC, Younis HS, Winzerling JJ. Biliary excretion of [(GS)(2)AsSe](-) after intravenous injection of rabbits with arsenite and selenate. Chem Res Toxicol. 2002 Nov;15(11):1466-71. doi: 10.1021/tx025538s. PMID 12437338
- [Background] Manley SA, George GN, Pickering IJ, Glass RS, Prenner EJ, Yamdagni R, Wu Q, Gailer J. The seleno bis(S-glutathionyl) arsinium ion is assembled in erythrocyte lysate. Chem Res Toxicol. 2006 Apr;19(4):601-7. doi: 10.1021/tx0503505. PMID 16608173
- [Background] Prince RC, Gailer J, Gunson DE, Turner RJ, George GN, Pickering IJ. Strong poison revisited. J Inorg Biochem. 2007 Nov;101(11-12):1891-3. doi: 10.1016/j.jinorgbio.2007.06.008. Epub 2007 Jun 13. PMID 17644180
- [Background] Carew MW, Leslie EM. Selenium-dependent and -independent transport of arsenic by the human multidrug resistance protein 2 (MRP2/ABCC2): implications for the mutual detoxification of arsenic and selenium. Carcinogenesis. 2010 Aug;31(8):1450-5. doi: 10.1093/carcin/bgq125. Epub 2010 Jun 27. PMID 20584751